CLINICAL TRIAL: NCT02052635
Title: A Phase IV, Randomised, Multi-Centre, Open Label Study, Comparing Ticagrelor Versus Clopidogrel in Non-ST Elevation Acute Coronary Syndrome (NSTE-ACS) Patients Undergoing Percutaneous Coronary Intervention (PCI) With Bivalirudin
Brief Title: Ticagrelor vs Clopidogrel in Non-ST Elevation Acute Coronary Syndrome Patients Undergoing PCI With Bivalirudin.
Acronym: NSTE-ACS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patient recruitment challenges, low enrolment, and a forecasted inability to complete the study in an acceptable timeframe
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5130L00065
Record Dates: First submitted 2014-01-14; First posted 2014-02-03 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Non-ST Elevation Acute Coronary Syndrome
Keywords: Percutaneous Coronary Intervention
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): 90 mg oral tablet
  Interventions: Drug: ticagrelor
- Clopidogrel (Active Comparator): 300 mg oral tablet
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: ticagrelor — Single loading dose of 180mg of ticagrelor at time of bivalirudin administration. Beginning 12 hrs following study drug administration, all pts in the ticagrelor arm will receive ticagrelor 90 mg (maintenance dose) approximately every 12 hrs until Follow-up telephone contact.
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: clopidogrel — Single loading oral dose of 600 mg of clopidogrel will be given at time of bivalirudin administration. Beginning 4 hrs following study drug administration, all pts in the clopidorgrel arm will receive ticagrelor 180 mg for the loading dose, followed by 90 mg maintenance dose approximately every 12 hours until the Follow-up telephone contact.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to determine if ticagrelor is as effective as clopidogrel in rate of onset and degree of platelet inhibition for patients with non-ST elevation of acute coronary syndrome (NSTE-ACS) undergoing ad hoc percutaneous coronary intervention (PCI) with bivalirudin.

DETAILED DESCRIPTION:
Multi-center, open-label study that will compare the onset of the platelet inhibition with ticagrelor versus clopidogrel when administered with bivalirudin during PCI on a background therapy of aspirin in patients with NSTE-ACS.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised for chest pain and potential acute coronary syndrome.
* Onset of the most recent cardiac ischemic symptoms must occur within 7 days before randomisation and documented by cardiac ischemic symptoms of ≥ 10 min duration at rest and at least 2 of the following: ST segment changes on electrocardiogram (ECG) indicative of ischemia, or Positive biomarker evdience of myocardial necrosis, or other risk factors such as: 60 yrs of age or older, previous myocardial infarction or coronary bypass surgery, multi-vessel coronary artery disease, diabetes mellitus, peripheral arterial disease, chronic renal disfunction.
* Females must be either surgically sterile or post-menopausal.
* Activated Clotting Time (ACT) </= 300 at the time of study treatment

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 30 days.
* Current acute complication of percutaneous coronary intervention or coronary bypass surgery.
* Any contraindication to ticagrelor, clopidogrel or bivalirudin.
* ST elevation myocardial infraction within 24 hours of study entry.
* Any indications for oral anticoagulation or aspirin dose other than 75 to 100 milligrams (mg) daily.
* Planned use of omeprazole or esomeprazole.
* Patients with known bleeding or coagulation disorders; patients requiring dialysis; patients who have an inability to swallow medication.
* Patients with known bleeding diathesis or coagulation disorder; history of intracranial bleed.
* Use of Intravenous (IV) heparin less than 2 hours before procedure.
* Sustained uncontrolled high blood pressure

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Cohen, MD, Principal Investigator — Newark Beth Israel Medical Center
Locations (8):
- United States (8):
  - Research Site, Jacksonville, Florida
  - Research Site, Lake Mary, Florida
  - Research Site, Macon, Georgia
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Rapid City, South Dakota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the USA. While 17 sites were activated, 9 sites enrolled patients, and only 7 sites successfully randomised patients. There were 34 patients screened, 21 screen failures and 13 randomised patients from 03 September 2014 and 20 April 2015. The study was terminated due to recruitment challenges and low enrolment concerns.
Groups:
- Ticagrelor: A single oral dose of 180 mg (90 mg tablet x2) of ticagrelor was administered at the time of the initial bivalirudin bolus administration.
- Clopidogrel: A single oral dose of 600 mg (300 mg tablet x2) of clopidogrel was administered at the time of the initial bivalirudin bolus administration.
Period: Overall Study
Arm/Group | Ticagrelor | Clopidogrel
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Clopidogrel | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (2.7) | 61.2 (14.7) | 62.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Units (PRU) Using VerifyNow™ at 0.5 Hours After Loading Dose
Description: PRU at 0.5 hours after a single oral loading dose of either ticagrelor 180 mg or clopidogrel 600 mg given at the time of the bivalirudin bolus
Time Frame: 0.5 hours post loading dose
Population: 10 patients were included in the pharmacodynamic (PD) analysis: 6 patients in the ticagrelor group and 4 patients in the clopidogrel group. 3 out 13 randomized pateints are excluded (1 patient without any PRU data, 2 pateints with protocol deviations)
Measure: Mean (Standard Deviation); unit: PRUs
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 6 | 4
PRUs | 289.2 (44.6) | 292.8 (38.7)

2. Primary Outcome: P2Y12 Reaction Units (PRU) Using VerifyNow™ at 1 Hour After Loading Dose
Description: PRU at 1 hour after a single oral loading dose of either ticagrelor 180 mg or clopidogrel 600 mg given at the time of the bivalirudin bolus
Time Frame: 1 hour post loading dose
Population: 10 patients were included in the PD analysis: 6 patients in the ticagrelor group and 4 patients in the clopidogrel group. Out of the 10 patients in the PD analysis, 1 patient in Ticagrelor group does not have PRU value at 1 hour post loading dose.
Measure: Mean (Standard Deviation); unit: PRUs
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 5 | 4
PRUs | 174.4 (88.9) | 249.8 (68.7)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) from informed consent to follow-up contact (4-7 days after treatment) and non-serious adverse events (AEs) of interest from time of randomisation to follow-up. All SAEs and non-serious AEs of interest will be recorded.
Description: This study just collects the following non-serious AEs of interest: bleeding events, dyspnoea, renal impairment/increased creatinine, brady arrhythmic event, increased liver function tests, gout/uric acid increases, pneumonia, gynecomastia, abnormal uterine bleeding, all malignancies excluding non-melanoma skin cancers.
Arm/Group | Ticagrelor | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 2/7 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=7) | Clopidogrel (N=6)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The target sample size for this study was 100 patients. But due to recruitment challenges and low enrolment,the study was terminated early with only 13 pateints randomized. No formal statistical analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall provide the Sponsor with copies of any materials at least thirty days in advance of publication, submission or presentation. At the request of the Sponsor, the PI shall withhold publication, submission for publication or presentation for a period of ninety days from the date on which the Sponsor receives the material to allow the Sponsor to take such measures as the Sponsor considers necessary to preserve its proprietary rights and/or protect its Confidential Information.